CLINICAL TRIAL: NCT01723761
Title: Correlations Between Arrhythmias, Climatic Variables and Air Pollution in Patients With Pacemaker and ICD, Followed by Remote Monitoring.
Brief Title: Correlations Between Arrhythmias and Air Pollution in Patients With Pacemaker and ICD
Acronym: ARIA
Status: Completed | Type: Observational
Sponsor: Effect Group, Italy (Network)
Responsible Party: Sponsor
Other Study IDs: ARIAPOL 01
Record Dates: First submitted 2012-10-23; First posted 2012-11-08 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Cardiac Arrhythmias
Keywords: air pollution; pacemaker; ICD; remote monitoring; supraventricular arrhythmias; ventricular arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is a clinical, observational study to evaluate the correlations among arrhythmias, climatic variables and air pollution in patients with pacemaker and implantable defibrillator (ICD), followed by remote monitoring.

Purpose of the Study: The purpose of this study is to test the hypothesis that changes in climatic variables, such as temperature, pressure and humidity, and changes of particulate matter <10µ (PM10), particulate matter <2.5µ (PM2.5), ozone (O3), carbon monoxide (CO), sulfur dioxide (SO2), nitrogen dioxide (NO2), are associated with an increase of supraventricular and ventricular arrhythmias.

Objectives: The aim of this study is to determine whether changes in variables conditions affect the electrical stability of the myocardium in patients with pacemakers and ICDs.

Population: male and female subjects, aged ≥ 18 years, implanted by a dual-chamber pacemaker, ICD or biventricular ICD (ICD-CRT). A total of 500 subjects from 15 cardiology centers of the Veneto region will be included.

DETAILED DESCRIPTION:
The primary objectives of this study are as follows:

* Determine if the changes of temperature, pressure and humidity, are associated with an increase of atrial and ventricular arrhythmias.
* Determine if the changes of air pollution (gas and particulate), are associated with an increase of atrial and ventricular arrhythmias.

The secondary objectives of the study are:

* Determine if the changes of air pollution (gas and particulate), are associated with significant changes in mean heart rate, rate variability rate and the percentage of paced beats.
* Determine whether changes in temperature, pressure or humidity, are associated with significant changes in mean heart rate, heart rate variability and the percentage of paced beats.
* Determine if the changes of temperature, pressure and humidity, are associated with an increase in mortality or hospitalization for myocardial infarction or congestive heart failure.
* Determine if the changes of air pollution (gas and particulate), are associated with an increase in mortality or hospitalization for myocardial infarction or congestive heart failure.

Study Design This is a prospective, observational study, which compares the occurrence of atrial and ventricular arrhythmias and changes in physiological parameters, with climatic variables and air pollution.

The study will include 500 subjects and will consist of two periods:

Screening: we will collect baseline characteristics of subjects in the clinical examination. The period recruitment will run for 12 months.

Follow-up: After written informed consent will be signed, subjects who meet the criteria for inclusion will be enrolled in the study and followed up for a minimum period of 12 months. The data obtained from the remote monitoring will be evaluated for the daily values provided for the parameters considered in the study.

Periodical visits in pacemaker clinic will be scheduled at the discretion of the referring cardiologist of the center. The arrhythmic events that will occur in this period, detected by means of remote monitoring or through other clinical evaluations will be recorded. Atrial arrythmias: atrial fibrillation or atrial flutter, supraventricular tachycardia.

Ventricular arrhythmias: ventricular tachycardia, ventricular fibrillation, ventricular extrasystoles.

Physiological variables: average heart rate (24 hours and at rest), heart rate variability, the percentage of paced beats.

In addition, any changes in drug therapies and all clinically relevant events, will be recorded.

During the same period data from monitoring stations of ARPAV (Regional Agency for Environmental Prevention and Protection of Veneto Region) will be collected.

Climatic variables: temperature, humidity, atmospheric pressure. Parameters of air pollution: PM10, PM2.5, O3, CO, SO2, NO2. For each patient, the data from the monitoring station ARPAV of the urban area of residence of the subject will be considered. The mean exposure level used in the analytical studies on the health effects is calculated on the average number of units active in the area. This number is usually of 2-3 units in large centers, while it is generally only 1 in small towns. The residents in centers without monitoring will be excluded from the study. The mean value is the best approximation ... to be continued page 6.

ELIGIBILITY:
Inclusion Criteria:

* Stable subjects,> 18 years, who have been implanted with a dual-chamber pacemaker, an ICD or ICD-CRT, compatible with remote monitoring systems, with daily transmission of data.

Exclusion Criteria:

* Presence of heart failure clinically manifest.
* Concomitant illness or a significant condition which severely limits the life expectancy.
* Any medical or surgical condition that, at the discretion of the investigator, places the patient at higher risk for his participation in the study.
* History of malignancy of any organ system in the last two years, whether treated or untreated, including leukemia and lymphoma (with the exception of basal cell carcinoma of the skin) if there is evidence of local recurrence of metastasis.
* History of drug or alcohol abuse in the last 2 years.
* Participation in another study of a drug or device within 30 days after randomization.
* Inability to communicate and to comply with all such obligations including the unwillingness or inability to give an informed consent.
* Residence in urban centers without environmental monitoring.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females, aged ≥ 18 years of age who have been implanted with a dual-chamber pacemaker, an ICD or ICD-CRT.
Sampling Method: Non-Probability Sample
Enrollment: 473 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
incidence of atrial arrhythmias. | 12- 24 months.
  The arrhythmic events that will occur during follow-up period, detected by remote monitoring or through other clinical evaluations, will be recorded and classified as follows: atrial fibrillation or atrial flutter, supraventricular tachycardia.
incidence of ventricular arrhythmias | 12-24 months
  The arrhythmic events that will occur during follow-up period, detected by remote monitoring or through other clinical evaluations, will be recorded and classified as follows: ventricular tachycardia, ventricular fibrillation, premature ventricular beats.

SECONDARY OUTCOMES:
Mean heart rate | 12-24 months
  Mean heart rate obtained by remote monitoring of pacemaker and ICDs.
Heart rate variability | 12-24 months
  Measures of heart rate variability calculated by devices and obtained by remote monitoring.
Percentage of paced beats | 12-24 months
  Percentage of paced beats will be measured by devices diagnostic and obtained via remote monitoring.
Mortality for myocardial infarction or heart failure. | 12-24 months
Hospitalization for myocardial infarction or heart failure. | 12-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Buja, MD, Principal Investigator — University of Padova
Locations (9):
- Italy (9):
  - Ospedale S.Maria dei Battuti - Cardiologia, Conegliano
  - Ospedale di ESte, Este
  - Mater Salutis, Legnago
  - Dell'Angelo Hospital, Mestre
  - Ospedale Civile, Mirano
  - Ospedale S. Valentino, Montebelluna
  - Dipartimento di Scienze Cardiologiche, Toraciche e Vascolari-Università di Padova, Padua
  - Civic Hospital, Portogruaro
  - Ospedale Ca' Foncello - Divisione di Cardiologia, Treviso

REFERENCES:
- [Derived] Folino F, Buja G, Zanotto G, Marras E, Allocca G, Vaccari D, Gasparini G, Bertaglia E, Zoppo F, Calzolari V, Suh RN, Ignatiuk B, Lanera C, Benassi A, Gregori D, Iliceto S. Association between air pollution and ventricular arrhythmias in high-risk patients (ARIA study): a multicentre longitudinal study. Lancet Planet Health. 2017 May;1(2):e58-e64. doi: 10.1016/S2542-5196(17)30020-7. Epub 2017 May 5. PMID 29851582